CLINICAL TRIAL: NCT06819046
Title: Improved Efficacy of Selective Laser Trabeculoplasty With the Addition of Rocklatan Post-treatment vs Artificial Tears Post-treatment
Status: Recruiting | Type: Observational
Sponsor: Colorado Ophthalmology Associates PC (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: KO-25-01
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Rocklatan: netarsudil and latanoprost ophthalmic solution 0.02%/0.005%
  Interventions: Drug: Rocklatan
- Systane Ultra: artificial tears
  Interventions: Drug: Systane Ultra

INTERVENTIONS:
Drug: Rocklatan — netarsudil and latanoprost ophthalmic solution 0.02%/0.005%
  Groups: Rocklatan
Drug: Systane Ultra — artificial tears
  Groups: Systane Ultra

SUMMARY:
A randomized, single-site, parallel-group, prospective study of patients who are candidates for SLT, to study the effect of IOP change with Rocklatan vs artificial tears.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Documented diagnosis of mild to moderate primary open angle glaucoma or ocular hypertension. Diagnosis of primary open angle glaucoma must be supported by the following:

  * 24-2 SITA faster within the last 6 months

    - With a mean deviation of 0 to -12 dB, excluding patients that meet severe criteria by having defects involving fixation or in two hemispheres.
  * OCT RNFL and optic nerve examination within the last 6 months

    * Diffuse or focal narrowing or notching of the optic disc rim, progressive narrowing of the neuroretinal rim, diffuse or localized thinning of the parapapillary RNFL, optic disc asymmetry of the two eyes consistent with loss of neural tissue, or thinning of the RNFL/GCA on examination or imaging
    * Progressive thinning on SD-OCT of 7 microns in inferior and superior quadrants or >4 micron loss in global RNFL thickness
    * Deviation from this ISNT rule (inferior, superior, nasal and temporal order of RNFL thickness with the inferior RNFL quadrant being the thickness)
* Candidate for bilateral SLT
* Post-washout, post-SLT IOPs between 28-10
* Gonioscopy findings of Schafer grade III and IV

Exclusion Criteria:

* Patients MD <-12, HVF defects in both hemispheres or involving fixation
* Medication conditions that prevent SLT
* Prior use of rho kinase inhibitor
* Previous SLT performed on either eye
* Prior MIGS implanted in either eye
* Prior or current intolerance of a Rho kinase inhibitor
* Uncontrolled IOP on maximum tolerated medical therapy; unable to washout
* Narrow angles or other angle abnormalities
* History of corneal disease or dystrophy, including endothelial dysfunction
* History of corneal edema
* Current or history of intra-ocular infection or inflammation
* History of retinal diseases that will could affect diagnostic testing
* Anticipated use of intra-ocular or topical steroids not associated with the study protocol
* Current participation of study drugs or devices or within 6 months prior to screening
* Pregnant or planning to be pregnant throughout the study
* Any condition in the opinion in the investigator that would potentially confound the results of this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients who are a candidate for bilateral SLT.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Mean diurnal IOP | 6 weeks of treatment

SECONDARY OUTCOMES:
Change in mean diurnal IOP from baseline | 28 days of treatment

OTHER OUTCOMES:
Percentage of patients who reach >20% IOP reduction from baseline | 6 weeks of treatment
Number of IOP spikes | 6 weeks of treatment
  IOP spike defined as IOP 50% above baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kingsley Okafor, MD, Principal Investigator — Colorado Ophthalmology Associates PC
Locations (1):
- Colorado Ophthalmology Associates PC, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No